CLINICAL TRIAL: NCT06520891
Title: "The Effect of The Combination Therapy of Statin and SGLT2i in The Treatment of Ischemic Heart Disease"
Status: Recruiting | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Abdelkader, "The Effect of The combination Therapy of Statin and SGLT2i in The Treatment of Ischemic Heart disease", Fayoum University
Other Study IDs: M716
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: 2 Drugs Are Statin and SGLT2i
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — collecting their blood samples and calculate the serum level of statin by using HPLC and calculate plasma level of SGLT2i by using HPLC as baseline first then after three months to predict the effect of each drug to another one, we will follow their cholesterol, triglyceride, low density lipo-protein and high density lipo-protein and we will also inspect their adverse effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients has ischemic heart failure: 30 patients will take statin.
  Interventions: Drug: Statin and SGLT2i
- Patients has ischemic heart: 30 patients will take both of statin and SGLT2i.
  Interventions: Drug: Statin and SGLT2i
- Patients has heart disease: 30 patients will take SGLT2i.
  Interventions: Drug: Statin and SGLT2i

INTERVENTIONS:
Drug: Statin and SGLT2i — Statin as atrovastatin SGLT2i as dapagliflozin

SUMMARY:
correlate the serum level of statin and SGLT2i when given as polytherapy with HPLC in ischemic heart failure patients and their laboratory tests (cholesterol, LDL, HDL and TG...)

DETAILED DESCRIPTION:
This is a prospective study that will carried out in Department of cardiology, Faculty of Medicine, Fayoum University during the period from 1 April 2024 to 1 Juley 2024. The study includes 90 Outpatients Clinic patients who met the inclusion criteria. Patients will provide written informed consent before involving in this study.

* we will split the 90 patients into three groups:

  1. 30 patients will take statin.
  2. 30 patients will take SGLT2i.
  3. 30 patients will take both of statin and SGLT2i.
* By collecting their blood samples and calculate the serum level of statin by using HPLC and calculate plasma level of SGLT2i by using HPLC as baseline first then after three months to predict the effect of each drug to another one, we will follow their cholesterol, triglyceride, low density lipo-protein and high density lipo-protein and we will also inspect their adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* we include patients established ischemic heart failure seen by a primary care provider to diagnose ischemic heart disease,
* They assessed the use of statin with SGLT2i.

Exclusion Criteria:

* We exclude patients with

  1. liver dysfunction.
  2. renal dysfunction.
  3. fungal infection.
  4. coagulation disorder.
  5. Pts using drugs that interact with SGLT2i.
  6. patients that will refuse to be enrolled in the Study or refuse to write informed consent.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the health care provider asks about patient's symptoms which may experience:
  * Chest pain, especially after physical exertion
  * Dizziness or fainting
  * Heart palpitations, which may feel like your heart fluttering or skipping beats
  * Shortness of breath
  * Swelling in your feet or ankles
    * brain natriuretic peptide (BNP) with 70% sensitivity and 99% specificity and N-terminal proBNP (NT-proBNP) with 99% sensitivity and 85% specificity which are Other HF-specific laboratory tests (especially in patients with a high possibility of heart failure) included. (18)
    * chest X-ray, transthoracic echocardiography (TTE), computerized tomography (CT) scans and magnetic resonance imaging (MRI) also other diagnostic tests for HF. (19)
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The Effect of The combination Therapy of Statin and SGLT2i in The Treatment of Ischemic Heart disease | Three months of follow up
  correlate the serum level of statin and SGLT2i when given as polytherapy with ECG in ischemic heart failure patients and their laboratory tests (cholesterol, LDL, HDL and TG...)

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa mohamed abdelkader, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
After ending the study, I will share it in magazin with other researchers